CLINICAL TRIAL: NCT02174289
Title: A Randomised Double-blinded Cross Over Study to Evaluate the Improvement of Left Ventricular Systolic Failure Using Targeted Left Ventricular Endocardial Lead Placement in Cardiac Resynchronisation Therapy.
Brief Title: LV Endocardial Cardiac Resynchronisation Therapy
Acronym: ENDO-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013PS003H; ISROTH20092 (Other Grant/Funding Number: Boston Scientific Global ISR program)
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiac Resynchronisation Therapy; Transseptal left ventricular endocardial lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Bi-ventricular Pacing (Active Comparator)
  Interventions: Device: Targeted left ventricular endocardial lead placement
- No Biventricular pacing (Placebo Comparator)
  Interventions: Device: Targeted left ventricular endocardial lead placement

INTERVENTIONS:
Device: Targeted left ventricular endocardial lead placement — The left ventricular endocardial lead will be passed through the intra-atrial septum

SUMMARY:
Cardiac resynchronisation therapy (CRT) is an established treatment for severe systolic heart failure with well documented benefits in symptom improvement and reduction of morbidity and mortality. However, upto 30% of patients do not respond to treatment despite fulfilling the recommended indications. Lack of clinical response may be the result of imperfect left ventricular lead placement in the veins around the heart with conventional techniques. Optimum lead placement may constrained by coronary venous anatomy and may overlie scarred heart muscle or may not be at the site of latest electrical depolarisation. In a further 10% of patients, conventional left ventricular lead placement is not possible for other technical reasons.

Left ventricular endocardial lead placement may overcome the limitations and allow placement to be guided by echocardiography, electrical mapping and the pattern of heart muscle scarring.

We aim to investigate if targeted left ventricular endocardial lead placement improves exercise capacity, heart failure symptoms, heart function and size, heart pumping efficiency and biochemical markers of heart strain. Each parameter will be assessed independently and as part of a composite cardiac performance score.

Patients with heart failure will be enrolled who require an endocardial left ventricular lead on clinical grounds as either conventional left ventricular lead implantation has technically failed or they have clinically non-responded to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* NYHA class II-IV
* LVEF ≤35%
* QRS ≥120 milliseconds
* Optimal tolerated medical therapy
* Either unable to position an LV lead via the standard coronary sinus on CRT implantation
* OR Recipient of a CRT-P or CRT-D system for greater than 6 months for standard indications AND limited improvement or worsened clinical status despite device optimisation
* Informed consent

Exclusion Criteria:

* Life-expectancy less than 1 year due to concomitant, non-cardiovascular disorders
* Previous atrial septal defect device closure.
* Chronic renal dialysis and End stage liver disease
* History of stroke, myocardial infarction, unstable angina, Coronary artery bypass grafting and coronary stenting within the last 3 months
* Presence of correctable valvular disease (aortic/mitral)
* Mitral valve prosthesis.
* Contra indication to vitamin K antagonist
* Unresolved intra-cardiac thrombus
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test | 3 months
  Improvement in peak oxygen consumption

SECONDARY OUTCOMES:
New NYHA Class | 3 months
  Change in New York Heart Association functional Class
6 minute walk | 3 months
  Change in 6 minute hall walk test distance
Quality of life | 3 months
  Minnesota Living with heart failure questionnaire score
Echocardiography | 3 months
  Change in size and function of the heart
Digital photoplethysmography | 3 months
  Cardiac output
Biochemical response | 3 months
  Change in eGFR (estimated glomerular filtration rate) and NT pro BNP (N terminal pro brain natriuretic peptide) levels.
Composite cardiac assessment score | 3 months
  Change in composite assessment score made up of symptom, exercise tolerance, echocardiographic and biochemical parameters.

OTHER OUTCOMES:
Freedom from adverse events | 1 year
  Acute: Tamponade, effusion, systemic thromboembolism; acute lead displacement and arrhythmia
  Chronic: systemic thromboembolism; lead displacement, disfunction or fracture; device related systemic infection; bleeding; arrhythmia
Medium term clinical outcomes | 6 months
  Assess medium term response to treatment with regards to symptoms, exercise tolerance, echocardiographic and biochemical parameters (as specified above), particularly systemic thrombosis.
Targeting success | Intra operative
  Success at targeting the site which produces the greatest haemodynamic response using echocardiogaphic speckle tracking, endocardial electrical mapping and myocardial perfusion scintigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wong, MD FESC, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Gras D, Bocker D, Lunati M, Wellens HJ, Calvert M, Freemantle N, Gervais R, Kappenberger L, Tavazzi L, Erdmann E, Cleland JG, Daubert JC; CARE-HF Study Steering Committee and Investigators. Implantation of cardiac resynchronization therapy systems in the CARE-HF trial: procedural success rate and safety. Europace. 2007 Jul;9(7):516-22. doi: 10.1093/europace/eum080. Epub 2007 May 31. PMID 17540662
- [Background] Jais P, Douard H, Shah DC, Barold S, Barat JL, Clementy J. Endocardial biventricular pacing. Pacing Clin Electrophysiol. 1998 Nov;21(11 Pt 1):2128-31. doi: 10.1111/j.1540-8159.1998.tb01133.x. PMID 9826866
- [Background] van Gelder BM, Scheffer MG, Meijer A, Bracke FA. Transseptal endocardial left ventricular pacing: an alternative technique for coronary sinus lead placement in cardiac resynchronization therapy. Heart Rhythm. 2007 Apr;4(4):454-60. doi: 10.1016/j.hrthm.2006.11.023. Epub 2006 Nov 29. PMID 17399634
- [Background] Nuta B, Lines I, MacIntyre I, Haywood GA. Biventricular ICD implant using endocardial LV lead placement from the left subclavian vein approach and transseptal puncture via the transfemoral route. Europace. 2007 Nov;9(11):1038-40. doi: 10.1093/europace/eum176. Epub 2007 Aug 17. PMID 17704095
- [Background] Jais P, Takahashi A, Garrigue S, Yamane T, Hocini M, Shah DC, Barold SS, Deisenhofer I, Haissaguerre M, Clementy J. Mid-term follow-up of endocardial biventricular pacing. Pacing Clin Electrophysiol. 2000 Nov;23(11 Pt 2):1744-7. doi: 10.1111/j.1540-8159.2000.tb07010.x. PMID 11139915
- [Background] Spragg DD, Dong J, Fetics BJ, Helm R, Marine JE, Cheng A, Henrikson CA, Kass DA, Berger RD. Optimal left ventricular endocardial pacing sites for cardiac resynchronization therapy in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2010 Aug 31;56(10):774-81. doi: 10.1016/j.jacc.2010.06.014. PMID 20797490
- [Background] Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18. doi: 10.1016/j.jacc.2011.12.030. Epub 2012 Mar 7. PMID 22405632
- [Background] Saba S, Marek J, Schwartzman D, Jain S, Adelstein E, White P, Oyenuga OA, Onishi T, Soman P, Gorcsan J 3rd. Echocardiography-guided left ventricular lead placement for cardiac resynchronization therapy: results of the Speckle Tracking Assisted Resynchronization Therapy for Electrode Region trial. Circ Heart Fail. 2013 May;6(3):427-34. doi: 10.1161/CIRCHEARTFAILURE.112.000078. Epub 2013 Mar 8. PMID 23476053